CLINICAL TRIAL: NCT03251807
Title: Effect of Low-Intensity Pulsed Ultrasound Applied on Temporomandibular Joint Region on Functional Treatment of Class II Malocclusion: A Randomized Controlled Trial
Brief Title: Effect of Low-Intensity Pulsed Ultrasound on Functional Treatment of Class II Malocclusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UDDS-Ortho-06-2017
Record Dates: First submitted 2017-08-13; First posted 2017-08-16 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Malocclusion, Angle Class II
Keywords: Low-intensity pulsed ultrasound; Twin-block; Functional treatment
MeSH Terms: conditions — Malocclusion, Angle Class II | interventions — Ultrasonic Waves

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Twin-block (Experimental): The patients in this control group will be treated using the Twin-block appliance.
  Interventions: Device: Twin-block
- Twin-block combined with LIPUS (Experimental): The patients in this experimental group will be treated using the Twin-block combined with LIPUS (Low-intensity pulsed ultrasound).
  Interventions: Device: Twin-block; Other: LIPUS (Low-intensity pulsed ultrasound)

INTERVENTIONS:
Device: Twin-block — Functional treatment will be achieved using the Twinblock appliance
Other: LIPUS (Low-intensity pulsed ultrasound) — Functional treatment will be combined with LIPUS (Low-intensity pulsed ultrasound )
  Arms: Twin-block combined with LIPUS

SUMMARY:
This experimental study will evaluate the effect of combined treatment with low-intensity pulsed ultrasound (LIPUS) and functional appliances (twin-block) on the correction of class II malocclusion, compared with the control group treated with functional appliances (twin-block) only.

The study sample will consist of 40 patients with class II malocclusion. The sample will be allocated randomly into two groups: control group and experimental group.

The functional appliance (twin-block) will be applied for all patients, while the low-intensity pulsed ultrasound (LIPUS) will be applied for the experimental group only. The skeleto-dental changes occurring after functional treatment will be assessed using cephalometric radiographs; pre and post- treatment changes for each group will be evaluated individually, and the two groups will be compared.

DETAILED DESCRIPTION:
Studies of the etiologic factors of Class II malocclusions recognize that most Class II malocclusions are a result of mandibular deficiency and not of maxillary excess. For many patients, especially adults, optimal overall results are best obtained using a combined orthodontic-surgical approach. However, treating such cases early while the patient is still growing, using mandibular propulsive functional appliances, can produce satisfactory improvement in the facial esthetics, and minimizes the need for surgical intervention in many cases.

Ultrasound (US), a form of mechanical energy that is transmitted through and into biological tissues as an acoustic pressure wave at frequencies above the limit of human hearing, is used widely in medicine as a therapeutic, operative and diagnostic tool. Therapeutic US, and some operative US. Previous studies on animals have found that therapeutic ultrasound (US) can stimulate and enhance mandibular growth when applied during the active growth period.

This study will evaluate the effect of low-intensity pulsed ultrasound (LIPUS) on the growth of mandible and the duration of functional treatment.

Twin-block will be applied to the two groups. While the control group will receive the twin-block only, the experimental group will receive the twin-block combined with low-intensity pulsed ultrasound (LIPUS) on Temporomandibular joint (TMJ) region.

Cephalometric radiographs will be obtained before and after functional treatment to evaluate the dento-skeletal changes.

ELIGIBILITY:
Inclusion Criteria:

* Angle class II malocclusion because of mandibular retrognathia
* O.J > 5 , SNB < 78
* Patient during growth spurt

Exclusion Criteria:

* TMJ disorders
* Poor oral hygiene
* Previous orthodontic treatment.
* Patients with syndromes, clefts, or craniofacial abnormalities.
* Reason of contraindication of functional treatment

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-10-12 (Actual); Study Completion 2019-03-12 (Actual)

PRIMARY OUTCOMES:
The duration of functional treatment | After functional treatment which will take approximately 8 months
  The duration of the functional treatment will be measured and compared between groups.

SECONDARY OUTCOMES:
Dentoskeletal effects of the functional treatment | Changes will be evaluated before and after functional treatment which will take approximately 8 months
  Dentoskeletal changes before and after functional treatment combined with Low-level Laser compared with those of the control group (SNA, SNB, ANB, Overjet ,…etc) using lateral cephalometric radiographs.

CONTACTS AND LOCATIONS:
Overall Officials: Ghiath Mahmood, PhD., Study Director — Department of Orthodontics, Faculty of Dentistry, Damascus University, Damascus, Syria
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No
The Individual participant data will be only available for the researchers in the department of Orthodontics, Damascus University

REFERENCES:
- [Background] El-Bialy T, El-Shamy I, Graber TM. Growth modification of the rabbit mandible using therapeutic ultrasound: is it possible to enhance functional appliance results? Angle Orthod. 2003 Dec;73(6):631-9. doi: 10.1043/0003-3219(2003)0732.0.CO;2. PMID 14719726
- [Background] El-Bialy T, Hassan A, Albaghdadi T, Fouad HA, Maimani AR. Growth modification of the mandible with ultrasound in baboons: a preliminary report. Am J Orthod Dentofacial Orthop. 2006 Oct;130(4):435.e7-14. doi: 10.1016/j.ajodo.2006.01.025. PMID 17045140
- [Background] Flores-Mir C, Major MP, Major PW. Soft tissue changes with fixed functional appliances in Class II division 1. Angle Orthod. 2006 Jul;76(4):712-20. doi: 10.1043/0003-3219(2006)076[0712:STCWFF]2.0.CO;2. PMID 16808582
- [Background] Jena AK, Duggal R, Parkash H. Skeletal and dentoalveolar effects of Twin-block and bionator appliances in the treatment of Class II malocclusion: a comparative study. Am J Orthod Dentofacial Orthop. 2006 Nov;130(5):594-602. doi: 10.1016/j.ajodo.2005.02.025. PMID 17110256
- [Background] Johns LD, Straub SJ, Howard SM. Analysis of effective radiating area, power, intensity, and field characteristics of ultrasound transducers. Arch Phys Med Rehabil. 2007 Jan;88(1):124-9. doi: 10.1016/j.apmr.2006.09.016. PMID 17207688
- [Background] Sun JS, Hong RC, Chang WH, Chen LT, Lin FH, Liu HC. In vitro effects of low-intensity ultrasound stimulation on the bone cells. J Biomed Mater Res. 2001 Dec 5;57(3):449-56. doi: 10.1002/1097-4636(20011205)57:33.0.co;2-0. PMID 11523040